CLINICAL TRIAL: NCT02359071
Title: Which Shift Characteristics Affect Handover Duration and Rates? A Prospective Multicentric Study
Brief Title: Shift Characteristics Affect Handover Duration and Rates.
Acronym: Handover
Status: Completed | Type: Observational
Sponsor: Ataturk University (Other)
Collaborators: Ankara Training and Research Hospital (Other); Duzce university-DUZCE (Unknown); Recep Tayyip Erdoğan University-RIZE (Unknown); Mustafa Kemal University (Other); DerinceTraining and Research Hospital- KOCAELI (Unknown); GATA Haydarpaşa Training Hospital, Istanbul (Other)
Responsible Party: Principal Investigator, Atıf, Atıf BAYRAMIGLU, Ataturk University
Other Study IDs: Atıf-001
Record Dates: First submitted 2015-02-04; First posted 2015-02-09 (Estimated); Last update posted 2015-11-20 (Estimated); Status verified 2015-02

CONDITIONS: Handover Duration
Keywords: handoff; signoff; handover; sign-out; shift change; Emergency Department
MeSH Terms: conditions — Emergencies

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Handovers with lower durations: equal or lower than 20 minutes
  Interventions: Other: handover duration, handover rate
- handovers with higher durations: Higher than 20 minutes
  Interventions: Other: handover duration, handover rate

INTERVENTIONS:
Other: handover duration, handover rate — To better analyze independent variables, we dichotomized the data. First, we dichotomized handover duration into two groups according to the median handoff time of 20 minutes. Second, we divided handover rates into two groups using the median rate of handovers per shift, which was 3.87%.

SUMMARY:
The primary aim of our study was to analyze the independent factors affecting handover duration in Emergency Department. The secondary aim was to identify the factors affecting Emergency Department handover rates.

DETAILED DESCRIPTION:
The primary aim in this study was to analyze the independent factors affecting handover duration in Emergency Department. Our secondary aim was to identify the factors affecting the Emergency Department handover rates. To better analyze independent variables, we dichotomized the data. First, we dichotomized handover duration into two groups according to the median handoff time of 20 minutes. Second, we divided handover rates into two groups using the median rate of handovers per shift, which was 3.87%.

ELIGIBILITY:
Inclusion Criteria:

The day and night shift handover , which are the interactive, verbal, bedside, and face-to-face interactions between the outgoing and incoming medical staff, were included.

Exclusion Criteria:

Handover locations other than bedside (n=3), handover methods except verbal communication (by paper (n=2)), and the use of information technology (n=1) were excluded to standardize the procedure.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: we obtained data streams from seven centers, and 267 completed records from different centre were included.
Sampling Method: Probability Sample
Enrollment: 267 (Actual)
Dates: Start 2013-09; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
the independent factors affecting handover duration in Emergency Department | 1-30 September 2013

SECONDARY OUTCOMES:
to identify the factors affecting Emergency Department handover rates. | 1-30 September 2013

CONTACTS AND LOCATIONS:
Overall Officials: Ali Karakus, Assoc. prof, Principal Investigator — Mustafa Kemal University; Ayhan Sarıtas, Assoc. prof, Principal Investigator — Duzce University; Gulhan Kurtoglu, specialist, Principal Investigator — Ankara Training and Research Hospital; Ozlem Bilir, Assist. Prof, Principal Investigator — Recep Tayyip Erdogan University; Ayhan Akoz, Assoc. prof., Principal Investigator — Ataturk University; Murat Eroglu, Assoc. prof, Principal Investigator — GATA Haydarpasa Military Hospital; Onur Karakayali, specialist, Principal Investigator — DerinceTraining and Research Hospital